CLINICAL TRIAL: NCT00263042
Title: Randomized, Multinational, Multicenter, Double-blind, Placebo-controlled, Two-arm Parallel Group Trial of Rimonabant 20 mg OD for Reducing the Risk of Major Cardiovascular Events in Abdominally Obese Patients With Clustering Risk Factors
Brief Title: Comprehensive Rimonabant Evaluation Study of Cardiovascular ENDpoints and Outcomes
Acronym: CRESCENDO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decision taken in light of demands by certain national health authorities
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC5826; 2005-002942-20 (EudraCT Number)
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-04

CONDITIONS: Cardiovascular Disease
Keywords: Myocardial infarction; cerebrovascular accident; obesity
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Stroke; Obesity | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rimonabant (Experimental): Rimonabant 20 mg once daily
  Interventions: Drug: Rimonabant
- Placebo (Placebo Comparator): Placebo (for Rimonabant) once daily.
  Interventions: Drug: Placebo (for Rimonabant)

INTERVENTIONS:
Drug: Rimonabant — Tablet, oral administration
  Other Names: SR141716; Acomplia
  Arms: Rimonabant
Drug: Placebo (for Rimonabant) — Tablet, oral administration
  Arms: Placebo

SUMMARY:
The primary objective is to show whether rimonabant reduces the risk of a heart attack (MI), stroke, or death from an MI or stroke in patients with abdominal obesity with other cardiovascular (CV) risk factors.

The secondary objective is to show whether rimonabant reduces the risk of MI, stroke, CV death, or CV hospitalization in these patients.

DETAILED DESCRIPTION:
The estimated study duration per patient is 36 to 53 months. All patients will be followed from randomization until a common study end date, which will occur when the last patient has been followed for 33 months.

ELIGIBILITY:
Inclusion Criteria:

Waist circumference >102 cm (40 inches) males, >88 cm (35 inches) females, with one coronary heart disease (CHD) equivalent or two major risk factors for cardiovascular disease.

* CHD equivalents:

  * Recent (within 3 years)documented heart attack
  * Documented symptomatic coronary artery disease
  * Recent (within 3 years) ischemic cerebrovascular episode (stroke or TIA)
  * Documented symptomatic peripheral arterial disease
* Major risk factors:

  * Documented type 2 diabetes mellitus
  * Metabolic syndrome (NCEP criteria)
  * Asymptomatic cerebrovascular, renal, or peripheral arterial disease, or past abdominal aortic aneurysm repair
  * Elevated high-sensitivity C-reactive protein
  * Age > or = 65 years for males, age > or = 70 years for females

Exclusion Criteria:

* Obesity of known endocrine origin
* Pregnant or breastfeeding women
* Very low calorie diet or weight loss surgery within past 6 months
* Presence of any severe medical or psychological condition that, in the opinion of the investigator, would compromise the patient's safe participation, including uncontrolled serious psychiatric illness
* Likely cardiovascular intervention within next 1 month
* Allergy to rimonabant or excipients, or prior participation in a rimonabant trial
* Receipt of investigational product within past 30 days

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18695 (Actual)
Dates: Start 2005-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
First occurrence of any of myocardial infarction, stroke or cardiovascular (CV) death | From randomization up to common study end date (33-50 months)

SECONDARY OUTCOMES:
First occurrence of any of myocardial infarction, stroke, CV death, and CV hospitalization | From randomization up to common study end date (33-50 months)
All-cause mortality | From randomization up to common study end date (33-50 months)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Topol, MD, Study Chair — Scripps Clinic; Deepak L. Bhatt, MD, Principal Investigator — The Cleveland Clinic
Locations (43):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- sanofi-aventis Australia & New Zealand administrative office, Macquarie Park, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Laval, Quebec, Canada
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Shangaï, China
- Sanofi-Aventis Administrative Office, Bogotá, Colombia
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Hong Kong, Hong Kong
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Dublin, Ireland
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Lysaker, Norway
- Sanofi-Aventis Administrative Office, Lima, Peru
- Sanofi-Aventis Administrative Office, Makati City, Philippines
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Madrid, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Bangkok, Thailand
- Sanofi-Aventis Administrative Office, Mégrine, Tunisia
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis Administrative Office, Guildford, United Kingdom

REFERENCES:
- [Result] Topol EJ, Bousser MG, Fox KA, Creager MA, Despres JP, Easton JD, Hamm CW, Montalescot G, Steg PG, Pearson TA, Cohen E, Gaudin C, Job B, Murphy JH, Bhatt DL; CRESCENDO Investigators. Rimonabant for prevention of cardiovascular events (CRESCENDO): a randomised, multicentre, placebo-controlled trial. Lancet. 2010 Aug 14;376(9740):517-23. doi: 10.1016/S0140-6736(10)60935-X. PMID 20709233
- [Derived] Bhatia G, Bansal V, Harismendy O, Schork NJ, Topol EJ, Frazer K, Bafna V. A covering method for detecting genetic associations between rare variants and common phenotypes. PLoS Comput Biol. 2010 Oct 14;6(10):e1000954. doi: 10.1371/journal.pcbi.1000954. PMID 20976246